CLINICAL TRIAL: NCT03414567
Title: Presence of Toxins from Smoking in the Follicular Fluid of Women with the Desire to Have Children Undergoing Intracytoplasmic Sperm Injection Treatment
Brief Title: Presence of Toxins from Smoking in the Follicular Fluid of Women Undergoing Intracytoplasmic Sperm Injection Treatment
Status: Completed | Type: Observational
Sponsor: Infertility Treatment Center Dortmund (Other)
Collaborators: TU Dortmund University (Unknown); Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Nicotine Folicular Fluid 2018
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Exposure to Toxins from Smoking; Female Infertility
Keywords: Follicular fluid; nicotine; cotinine; Benzo(a)pyrene
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Follicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Non-smoker
- Study Group: Smoker

SUMMARY:
Smoking is associated with many adverse health effects like circulatory disorders, pulmonary diseases or heart diseases. It was also shown that smoking correlates with a significantly higher risk for miscarriage, preterm birth or a significantly decreased implantation rate or life birth rate, thus affects the chance to have children.

Combustion of tobacco products results in more than 4.000 toxic and/or carcinogenic substances. Examples of such substances are the carcinogenic substance Benzo(a)pyrene or nicotine and its main degradation product cotinine. Although the adverse effects of these substances were analyzed in many biological systems (e.g. cell culture, mouse model systems), less is known about the bio-accumulation in human tissue, especially in ovarian tissue or the follicular fluid (FF).

The aim of this study is therefore to analyze the bio-accumulation of nicotine, cotinine and Benzo(a)pyrene in the follicular fluid of women with the unfulfilled desire to have children undergoing an intracytoplasmic sperm injection (ICSI) treatment. The analysis will be performed using a sensitive gas chromatography-mass spectroscopy (GC) in a control group (non-smoker) and a study group (smoker). For each group, a correlation analysis between the amount of toxic and/or carcinogenic substances and the clinical outcome (e.g. clinical pregnancy rate, fertilization rate) will be performed. In combination with a patient questionnaire, it will be possible to analyze the risk of smoking, the bio-accumulation of toxic substances in the follicular fluid, and the chance to have children.

DETAILED DESCRIPTION:
The desire to have children can be influenced by a number of factors. Besides hormonal factors, age and body weight, or genetic disorders, smoking may play an important role. It was shown that cigarette smoking correlates with a significantly decreased implantation and life birth rate, and a significantly higher risk for miscarriage or preterm birth. Moreover, limitations of the oocyte quality, a decreased thickness of the Zona Pellucida, or spindle disorders were reported. Overall, smokers are much less likely to succeed in pregnancy as published by the American Society for Reproductive Medicine (ASRM) in 2012. Although general tobacco consumption in Germany is declining, about 30% of women of childbearing age (between 18 and 45 years) smoke (German Federal Office of Statistics, 2013).

Combustion of tobacco products (and additives like glycerin, menthol or sorbic acid) results in the formation of more than 4.000 toxic and/or carcinogenic substances. Two of these substances are nicotine and its main degradation product cotinine, another example is the carcinogenic substance Benzo(a)pyrene. The nicotine clearance in the human body is relatively fast - the half-life of nicotine is less than 2 hours in the human body. However, cotinine with a half-life of more than 16 hours is an appropriate biomarker to study the bio-accumulation of nicotine/cotinine. The effect of nicotine, cotinine or Benzo(a)pyrene on the reproductive system has already been investigated in various animal model systems and some clinical trials. For example, nicotine limits progesterone and estrogen biosynthesis, reduces peripheral blood flow, and reduces contractility of the fallopian tubes and uterus. Benzo(a)pyrene impairs cell proliferation as well as estrogen biosynthesis. It has also been implicated in DNA damaging mechanisms.

Nevertheless, little is known about the bio-accumulation of these toxic substances in human tissue, especially in the reproductive system (e.g. ovarian tissue or the follicular fluid). Some published studies were additionally limited because of their limited sample size (n<50) or non-sensitive analyzing tools (e.g. enzyme-linked immunosorbent assay (ELISA) analysis). The aim of this study is therefore to analyze the bio-accumulation of nicotine, cotinine and Benzo(a)pyrene in the follicular fluid of women with the unfulfilled desire to have children undergoing an intracytoplasmic sperm injection treatment using an ultra-sensitive gas chromatography-mass spectroscopy in a control group (non-smoker) and a study group (smoker). For each group, a sample size of n=150 will be included. This makes it possible to perform a statistical analysis regarding the presence of smoking pollutants in the follicular fluid and the associated clinical parameters (e.g. clinical pregnancy outcome, oocyte count, fertilization rate) between the study and control group. In combination with a patient questionnaire, it will be possible to identify the risk of smoking, the bio-accumulation of toxic substances in the follicular fluid and the desire to have children.

ELIGIBILITY:
Inclusion Criteria:

- healthy females without sterility factors

Exclusion Criteria:

* Endometriosis
* Polycystic ovary syndrome (PCO)
* Neoplasia (ovary, Uterus, breast)
* Anti-Müllerian hormone (AMH) <1 ng/ml

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female patients seeking ICSI treatment because of male subfertility
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 28 days after ICSI treatment
  Presence of amniotic cavity and heartbeat after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Dieterle, MD, Principal Investigator — Infertility Treatment Center Dortmund
Locations (1):
- Infertility treatment center Dortmund, Dortmund, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trapphoff T, Ontrup C, Krug S, Dieterle S. Consumption of hookahs, e-cigarettes, and classic cigarettes and the impact on medically assisted reproduction treatment. Sci Rep. 2024 Apr 26;14(1):9597. doi: 10.1038/s41598-024-60251-y. PMID 38671174
- See also: Trapphoff et al., 2024 (Consumption of hookahs, e-cigarettes, and classic cigarettes and the impact on medically assisted reproduction treatment) — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC11053167/